CLINICAL TRIAL: NCT06852144
Title: Ruolo Della PET/TC Nella Valutazione di Patologia Tiroidea in un Centro di Medicina Nucleare ad Alto Volume Diagnostico
Brief Title: PET-TC in Thyroid Evaluation
Acronym: PEPATI-MN-2024
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PEPATI-MN-2024; 322/2024/Oss/AOUBo (Registry Identifier: AOU Bologna)
Record Dates: First submitted 2025-02-11; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-12

CONDITIONS: Medullary Thyroid Carcinoma; Hyperparathyroidism; Parathyroid Carcinoma
Keywords: PET/TC; 18F/FDG; hyperparathyroidism
MeSH Terms: conditions — Carcinoma, Medullary; Hyperparathyroidism; Parathyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pepati group: Patients belonging to the U.O. of Nuclear Medicine IRCCS - University Hospital of Bologna - Polyclinic S. Orsola, who have performed or are to perform PET/CT for thyroid/parathyroid disease or other clinical indication with incidental detection of thyroid/parathyroid disease or patients undergoing PET/CT with known thyroid/parathyroid disease (for example, patients with thyroid nodules already subjected to needle aspiration) as part of the normal care path for a period of 5 years and 6 months.
  Interventions: Other: clinical practice drug treatment

INTERVENTIONS:
Other: clinical practice drug treatment — Observational, prospective and retrospective study, transversal, non-profit, monocentric. All data of patients affected/ afferents to theU.O. of Nuclear Medicine of the IRCCS AOU of Bologna will be collected submitted/ who will undergo a PET/ CT investigation for thyroid pathology or other indication with incidental feedback of thyroid uptake and patients who have They undergo PET/CT with known thyroid disease. Of these patients will be collected the personal data, clinical news, data related to PET/ CT (dedicated software e.g. MIM), biochemical/ laboratory and anatomopathological (for operated patients), any other imaging investigations already performed and to be performed later by normal clinical practice. The medical nuclear images will be evaluated by at least two nuclear medical experts, with qualitative, semi-quantitative and radiometric parameters as far as possible. Patients will be treated according to normal clinical practice.

SUMMARY:
The thyroid gland may have a diffuse or focal uptake of numerous PET/CT radiopharmaceuticals and this may be correlated with underlying benign and malignant thyroid/parathyroid pathologies.

It is not clear at present if the uptake of the radiopharmaceutical alone is associated with a potential malignancy of the disease.

The aim of the study is to collect evidence and consolidate the diagnostic power of PET/CT, to identify any predictive parameters that can determine whether PET positivity/negativity can in the future avoid unnecessary tests such as needle aspiration.

DETAILED DESCRIPTION:
The primary objective of the study is to measure the diagnostic performance of PET/CT (with tracers used in our Center for Nuclear Medicine by normal clinical practice), in the identification of malignancy of thyroid or parathyroid findings, compared to cytological/histological examination in patients with known thyroid and/or parathyroid disease or in patients with incidental findings. The secondary objective is to find functional parameters and predictive imaging of malignancy/benign and risk class of the lesion.

ELIGIBILITY:
Inclusion Criteria:

For the retrospective part:

* Patients aged >18 years,
* Findings of hypercaptant of thyroid/parathyroid relevance to PET/CT or known thyroid or parathyroid pathology and subsequent execution of PET/CT according to normal clinical practice,
* Patients with cytological examination derived from needle aspiration performed no more than 12 months time apart from PET/CT.
* Obtaining informed consent

For the prospective part:

* Patients aged >18 years,
* Finding hypercaptant findings of thyroid/parathyroid relevance to PET/CT or known thyroid or parathyroid pathology and subsequent execution of PET/CT according to normal clinical practice.
* Patients scheduled for agesult to be no more than 12 months.
* Obtaining informed consent

Exclusion Criteria:

* Nothing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients belonging to the U.O. of Nuclear Medicine IRCCS - University Hospital of Bologna - Polyclinic S. Orsola, who have performed or are to perform PET/CT for thyroid/parathyroid disease or other clinical indication with incidental detection of thyroid/parathyroid disease or patients undergoing PET/CT with known thyroid/parathyroid disease (for example, patients with thyroid nodules already subjected to needle aspiration) as part of the normal care path for a period of 5 years and 6 months.
Sampling Method: Probability Sample
Enrollment: 418 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance | 5 years and 6 months
  Sensitivity, specificity, AUC, detection rate, accuracy, positive and negative predictive value compared to the reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine, IRCCS, Azienda Ospedalierio-Universitaria di Bologna, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cocchiara G, Fazzotta S, Palumbo VD, Damiano G, Cajozzo M, Maione C, Buscemi S, Spinelli G, Ficarella S, Maffongelli A, Caternicchia F, Ignazio Lo Monte A, Buscemi G. The medical and surgical treatment in secondary and tertiary hyperparathyroidism. Review. Clin Ter. 2017 Mar-Apr;168(2):e158-e167. doi: 10.7417/CT.2017.1999. PMID 28383630
- [Result] Bertagna F, Albano D, Giovanella L, Giubbini R, Treglia G. F18-choline/C11-choline PET/CT thyroid incidentalomas. Endocrine. 2019 May;64(2):203-208. doi: 10.1007/s12020-019-01841-z. Epub 2019 Jan 12. PMID 30637562
- [Result] Marcus C, Whitworth PW, Surasi DS, Pai SI, Subramaniam RM. PET/CT in the management of thyroid cancers. AJR Am J Roentgenol. 2014 Jun;202(6):1316-29. doi: 10.2214/AJR.13.11673. PMID 24848831